CLINICAL TRIAL: NCT03560401
Title: Is Postoperative Bracing Necessary After Spine Surgery for Degenerative Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2015-08-006ACF
Record Dates: First submitted 2017-12-21; First posted 2018-06-18 (Actual); Last update posted 2018-06-18 (Actual); Status verified 2018-06

CONDITIONS: Degenerative Lumbar Spinal Stenosis; Lumbarsacral Orthosis; Transforaminal Lumbar Interbody Fusion
Keywords: Bracing; transforaminal lumbar interbody fusion (TLIF); outcome; fusion rate
MeSH Terms: interventions — Braces

STUDY DESIGN:
Intervention Model Description: Patients in the brace group were instructed to wear a rigid brace (Knight-Taylor [chairback] brace) full-time for 12 weeks, except when bathing or lying in bed. Patients in the no brace group were instructed to wear a soft corset for 2 weeks, after which it was weaned off. All patients started wearing the brace or corset during their first ambulation out of bed following drainage tube removal after the surgery.
Who Masked: Investigator
Masking Description: Patients eligible for the study were selected by an independent research assistant. The study was explained, and informed consent was obtained from patients before the surgery. Using a randomization sequence, the patients were assigned to the brace or no brace group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brace group (Experimental): After spinal surgery, patients in the brace group were instructed to wear a rigid brace (Knight-Taylor [chairback] brace) full-time for 12 weeks, except when bathing or lying in bed.
  Interventions: Device: Knight-Taylor [chairback] brace
- No brace group (No Intervention): After spinal surgery, patients in the no brace group were instructed to wear a soft corset for 2 weeks, after which it was weaned off.

INTERVENTIONS:
Device: Knight-Taylor [chairback] brace — Knight-Taylor [chairback] brace, is one kind of rigid lumbosacral orthosis. The manufacturer was Rehabilitation and Technical Aid Center, Taipei Veterans General Hospital.
  Arms: Brace group

SUMMARY:
This study was started from Oct. 2015. This study aimed to evaluate the outcome of bracing following transforaminal lumbar interbody fusion (TLIF) in patients with degenerative lumbar spine diseases.

DETAILED DESCRIPTION:
The inclusion criteria were age older than 18 years and undergoing TLIF for degenerative lumbar disc disease, spinal stenosis, or spondylolisthesis. Those who had spinal fracture, spinal infection, spinal tumor, and a history of previous spinal surgery; and those who were lost to follow-up or failed to complete the questionnaires were excluded.

Patients eligible for the study were selected by an independent research assistant. The study was explained, and informed consent was obtained from patients before the surgery. Using a randomization sequence, the patients were assigned to the brace or no brace group. The attending surgeons and patients were blinded before the surgery.

Patients in the brace group were instructed to wear a rigid brace (Knight-Taylor [chairback] brace) full-time for 12 weeks, except when bathing or lying in bed. Patients in the no brace group were instructed to wear a soft corset for 2 weeks, after which it was weaned off. All patients started wearing the brace or corset during their first ambulation out of bed following drainage tube removal after the surgery.

The success of interbody fusion was evaluated by computed tomography (CT) at the 6-month postoperative follow-up using the Brantigan-Steffee-Fraser (BSF) classification6. Radiographic fusion (BSF-3) was defined as bone bridging at least half of the fusion area with at least the density originally achieved at surgery. Radiographic locked pseudarthrosis (BSF-2) was indicated by lucency visible in the middle of the cage with solid bone growing into the cage from each vertebral end plate. Radiographic pseudarthrosis (BSF-1) was indicated by collapse of the construct, loss of disk height, vertebral slip, broken screws, displacement of the cage, significant resorption of the bone graft, or lucency visible around the periphery of the graft or cage.

Perioperative complications, such as wound infection, epidural hematoma, intraoperative dural tear, nerve root damage, and implant dislodgement, were recorded, as were the reoperations and medically related complications within 6 months. The implant-related complications, such as screw loosening, cage migration, or broken screws, detected using plain radiograph at each follow-up and CT scan at the latest follow-up were also recorded. Pedicle screw loosening was defined as a radiolucent zone around the screw on a CT scan at the 6-month follow-up

Statistical analysis was performed using SPSS (version 22.0, IBM Corp., Armonk, NY, USA). Categorical data were compared using chi-square or Fisher's exact test. Continuous data were compared using the independent t-test. The two-tailed significance level was set at p <0.05.

ELIGIBILITY:
Inclusion Criteria:

* Patients underwent TLIF for degenerative lumbar disc disease, spinal stenosis, or spondylolisthesis

Exclusion Criteria:

* spinal fracture, spinal infection, spinal tumor, and a history of previous spinal surgery; and those who were lost to follow-up or failed to complete the questionnaires

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2015-10-20 (Actual); Primary Completion 2016-12-25 (Actual); Study Completion 2017-10-22 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale and Oswestry Disability Index functional outcome | 6 months of postoperative follow-up
  Visual Analogue Scale score was patient reported pain scale. The 0 score is no any pain. THe 10 score is the most pain ever. THe more the score the worsen the pain .
  The Oswestry Disability Index score is the most common used score for lumbar spine disability score. This score had only 10 questions, and all of the questions are related to pain and daily activity. 0 score is no any disability or pain. 100 score is the worst.

SECONDARY OUTCOMES:
interbody fusion rate | postoperative 6 months follow-up
  use CT scan to evaluate the bone union condition after interbody fusion of lumbar spine
complication | postoperative 6 months follow-up
  any undesirable condition after spinal surgery
reoperation | postoperative 6 months follow-up
  any reoperation after primary spinal surgery

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Chau Chang, M.D, Study Director — Taipei Veterans General Hospital, Taiwan
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Yee AJ, Yoo JU, Marsolais EB, Carlson G, Poe-Kochert C, Bohlman HH, Emery SE. Use of a postoperative lumbar corset after lumbar spinal arthrodesis for degenerative conditions of the spine. A prospective randomized trial. J Bone Joint Surg Am. 2008 Oct;90(10):2062-8. doi: 10.2106/JBJS.G.01093. PMID 18829902
- [Result] Soliman HAG, Barchi S, Parent S, Maurais G, Jodoin A, Mac-Thiong JM. Early Impact of Postoperative Bracing on Pain and Quality of Life After Posterior Instrumented Fusion for Lumbar Degenerative Conditions: A Randomized Trial. Spine (Phila Pa 1976). 2018 Feb 1;43(3):155-160. doi: 10.1097/BRS.0000000000002292. PMID 28632643